CLINICAL TRIAL: NCT00904046
Title: Pathophysiology of Uric Acid Nephrolithiasis
Acronym: IUAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Khashayar Sakhaee, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Study00000125; 1R01DK081423 (NIH)
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Uric Acid Kidney Stone Disease
Keywords: Uric acid; Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Pioglitazone; 2,4-thiazolidinedione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental): For 60 Aim 2 Subjects Only - Pioglitazone (Actos)
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): For 60 Subjects in Aim 2 Only - Placebo for Pioglitazone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 30 mg orally daily for 6 months
  Other Names: Thiazolidinedione
  Arms: Pioglitazone
Drug: Placebo — Placebo taken orally once a day for 6 months.
  Arms: Placebo

SUMMARY:
This study has two aims:

Aim 1: To determine the presence of accumulation of fat within cells and the functional consequences of this in the kidney by correlating kidney fat content with urine test results.

Aim 2: The investigators will evaluate the effect of thiazolidinedione (pioglitazone) on excess fatty acid accumulation in kidney tissue and its correlation with uric acid stone formation in subjects with uric acid stones.

Pioglitazone is already U.S. Food & Drug Administration (FDA)-approved for the treatment of type 2 diabetes, but is not approved by the FDA for treating or preventing or diagnosing stone risk.

DETAILED DESCRIPTION:
The study will use a combination of cell culture, animal, and human studies employing some of the latest technologies in magnetic resonance spectroscopy and single-photon emission computed tomography, combined with classical physiology, biochemistry, and molecular biology to test four interrelated hypotheses. There is increased uptake of free fatty acids into the kidney as a result of higher circulating levels as well as preferential transport by the proximal tubule as part of a "conditioning" effect. The increased provision of free fatty acid supplies metabolic substrate for ATP generation hence reducing the consumption of other substrates such as glutamine, which is the principal source of ammoniagenesis by the proximal tubule. This substrate competition, or metabolic switch, can lower the formation of the major urinary buffer ammonia, even in the absence of injury to the proximal tubule. With sustained lipid loading of the proximal tubule that exceeds its oxidative capacity, lipid storage is first activated but with time, toxic lipid metabolites may build up. We have evidence that excess saturated fat, which is prevalent in the Western diet, leads to proximal tubule lipotoxicity manifested as endoplasmic reticulum (ER) leakage/stress, and we propose that defective ammoniagenesis is part of a broader lipotoxic phenotype. We further propose that accumulation of a specific lipid species may be responsible for the toxicity. To test whether proximal tubule steatosis and lipotoxicity in humans have a functional consequence, we will study uric acid stone formers. Having previously shown that thiazolidinediones (TZD) reduce renal steatosis and lipotoxicity and improve ammonium excretion in animals, we have initiated a randomized intervention trial with TZD or placebo in human uric acid stone formers. The interim analysis showed that after 6 months of TZD therapy, stone formers had improved urinary biochemical parameters and reduced propensity for uric acid precipitation. We will continue this trial but add a novel highly sensitive method to non-invasively measure renal fat, testing whether improvement in urinary biochemistry associates with reduction of renal fat. This proposal addresses fundamental concepts of renal tubular lipid biology and lipotoxicity, and clinically will shift the paradigm of uric acid stone therapy from empiric urinary alkalinization to specific reduction in renal fat. We will also introduce cutting-edge human imaging studies for kidney research.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with uric acid kidney stone disease
* Age > 21 years

Exclusion Criteria:

* Body weight> 350 lb
* Chronic alcohol use
* Chronic liver disease
* Chronic renal disease
* Anemia
* Contraindication to pioglitazone use:

  * history of congestive heart failure NYHA class III or IV
  * significant pedal edema
  * liver failure
  * not willing to practice an effective contraception for the duration of the study
* Thiazolidinedione use in the preceding 18 months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-01-15 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Reversal of renal lipotoxicity will occur with pioglitazone. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Khashayar Sakhaee, MD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center - Center for Mineral Metabolism, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Mineral Metabolism Website — https://www.utsouthwestern.edu/education/medical-school/departments/min-metab-center/research.html